CLINICAL TRIAL: NCT03239847
Title: Cost Effectiveness of the EndoPhys Pressure Sensing Access System vs. Radial A-line for Intra-operative Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Froehler, Asst. Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 160877
Record Dates: First submitted 2017-07-21; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Anesthesia team will not be made aware of the purpose of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoPhys Sheath and Radial Arterial Line (Experimental): This group of patients will have both the EndoPhys sheath and the radial arterial line placed during surgery.
  Interventions: Other: EndoPhys Sheath and Radial Arterial Line
- EndoPhys Sheath (Experimental): This group of patients will only receive the EndoPhys sheath during surgery.
  Interventions: Other: EndoPhys Sheath

INTERVENTIONS:
Other: EndoPhys Sheath and Radial Arterial Line
  Arms: EndoPhys Sheath and Radial Arterial Line
Other: EndoPhys Sheath
  Arms: EndoPhys Sheath

SUMMARY:
This study aims to compare the time difference between radial arterial line placement and use of the EndoPhys sheath, as well as, assess the cost effectiveness of the EnoPhys sheath vs. use of a radial arterial line based on device and operating room costs.

ELIGIBILITY:
Inclusion Criteria:

* All elective neuro endovascular procedures requiring general anesthesia and continuous invasive blood pressure monitoring
* Adequate access to both the radial or femoral artery

Exclusion Criteria:

* Pre-operative identification of contra-indication for radial arterial line placement
* Hemodynamic instability
* Need for continued post-operative invasive blood pressure monitoring
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Total Cost | Patient time in operating room (approximately 2 hours)
  Total cost of each approach, as defined by the sum of material (device) costs plus the value of operative room time per minute.

SECONDARY OUTCOMES:
Difference in preparation time between the two approaches | From onset of anesthesia to successful insertion of the catheter (approximately 30 minutes)
Complication rates between the two groups. | Patient time in operating room (approximately 2 hours)
Associated anticipated costs of complications between the two groups. | Patient time in operating room (approximately 2 hours)
Patient satisfaction as assessed by post-operative questionnaire | Questionnaire is assessed post-operatively at one day and at the 2-4 week follow up (approximately 5 minutes to assess)
Anesthesiologist satisfaction as assessed by post-operative questionnaire | Questionnaire is assessed post-operatively in the operating room (approximately 5 minutes to assess)
Technical success of EndoPhys sheath for blood pressure measurement and accuracy as compared to the radial arterial line. | Upon EndoPhys sheath insertion until it is removed from the femoral artery (approximately 1.5 hours)
Sensitivity analysis to evaluated variation in times for arterial line placement | From onset of anesthesia to successful insertion of the catheter (approximately 30 minutes)
Sensitivity analysis to evaluated variable operating room time costs | Patient time in operating room (approximately 2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Froehler, MD, PhD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Froehler MT, Chitale R, Magarik JA, Fusco MR. Comparison of a pressure-sensing sheath and radial arterial line for intraoperative blood pressure monitoring in neurointerventional procedures. J Neurointerv Surg. 2018 Aug;10(8):784-787. doi: 10.1136/neurintsurg-2018-013769. Epub 2018 Feb 27. PMID 29487193